CLINICAL TRIAL: NCT05191082
Title: Manufacturing, Characterization and Evaluation of the Effect of Silk Fibroin Membranes, Loaded or Not With Neurotensins on Open Wounds in the Palate: Randomized Clinical Study
Brief Title: Manufacturing, Characterization and Evaluation of the Effect of Silk Fibroin Membranes, Loaded or Not With Neurotensins on Open Wounds in the Palate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEPJMF 12
Record Dates: First submitted 2021-12-23; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Wound Healing; Palate; Wound
Keywords: Periodontology; Wound healing; Silk fibroin; Randomized clinical trial; Drug Delivery System
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel, superiority, randomized clinical trial with a 3 months of follow-up
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (Sham Comparator): The palatal wound area will not receive any treatment
  Interventions: Procedure: Palatal Wound
- Silk Fibroin Film - SF (Experimental): The palatal wound area will receive silk fibroin film as a dressing
  Interventions: Procedure: Palatal Wound; Device: Palatal Wound treated with Silk Fibroin Film
- Neurotensin-loaded Silk Fibroin Film - SF + NT (Experimental): The palatal wound area will receive a neurotensin-loaded silk fibroin film as a drug delivery system
  Interventions: Procedure: Palatal Wound; Device: Palatal Wound treated with Neurotensin-loaded Silk Fibroin Film

INTERVENTIONS:
Procedure: Palatal Wound — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive 4.0 silk sutures.
Device: Palatal Wound treated with Silk Fibroin Film — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive a silk fibroin film and 4.0 silk sutures.
  Arms: Silk Fibroin Film - SF
Device: Palatal Wound treated with Neurotensin-loaded Silk Fibroin Film — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive a silk fibroin film loaded with neurotensin and 4.0 silk sutures.
  Arms: Neurotensin-loaded Silk Fibroin Film - SF + NT

SUMMARY:
The aim of the present study will be to manufacture and characterize silk fibroin membranes loaded or not with neurotensin and to evaluate clinical, patient-centered and immunological parameters the effect of using these membranes on open wounds on the human palate.

DETAILED DESCRIPTION:
Surgical procedures for the reconstruction of gingival and peri-Implant tissues with the purpose of restoring function and aesthetics are commonly used in the dental practice. The use of free gingival graft (FGG), despite being considered the gold standard, causes great morbidity and postoperative pain. Thus, in order to reduce these complications, some biomaterials have been explored to accelerate healing and bring greater comfort to the patient. The present study aims to: 1. manufacture silk fibroin membranes (SF), loaded or not with neurotensin (NT); 2. evaluate, clinically and immunologically, the effect of the membranes on open wounds at palate sites. After the manufacture of the membranes they will be characterized by visual aspect, thickness, mechanical properties, surface texture, water vapor permeability, enzymatic degradation and swelling. Posteriorly, sixty six (n = 66) patients requiring exodontia and ridge preservation for future implant placement will be randomly assigned into three groups: Control - Free Gingival Graft (n = 22): extraction and Free Gingival Graft for sealing the alveolus entrance; Group SF - Fibroin membrane (n = 22): extraction and Free Gingival Graft for sealing the alveolus entrance and placement of the fibroin membrane at the palatal wound site; Group SF + NT - Free Gingival Graft + Neurotensin-loaded Fibroin Membrane (n = 22): extraction and Free Gingival Graft for sealing the alveolus entrance and placement of neurotensin-loaded fibroin membrane at the palatal wound site. The repair of the palatine donor area will be evaluated by clinical parameters such as remaining wound area, tissue thickness, re-epithelialization and early-wound healing index at baseline, 7, 14, 21, 30, 45, and 90 days after the procedure; and patient-centered outcomes by post-operative discomfort, tissue edema and number of analgesic pills used for 14 days after the procedure. In addition, inflammatory cytokines and growth factors will be assessed using the palatal wound inflammatory exudate 3 and 7 days after surgery. For the descriptive statistics, the mean ± standard deviation will be used; Normality: Shapiro-Wilk test; Clinical trials: ANOVA for intra and inter group calculations + Tukey test for multiple comparisons when the Shapiro-Wilk p value ≥ 0.05. If p Shapiro-Wilk <0.05, will be analyzed using the Friedman test (intragroup) and Mann-Whitney tests (intergroup); Parameters centered on patients: T test.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old, healthy systemically, with good oral hygiene, assessed by means of a plaque index and gingival index less than 25% (O'Leary et al., 1972)
* Patients with no morphological or pathological changes in the donor palatal region;
* Patients who have an indication for extraction and with an indication to preserve the socket for future implant installation;
* The tooth included in the study, as well as the adjacent teeth, must not have loss of periodontal insertion.

Exclusion Criteria:

* Patients with systemic problems (cardiovascular changes, blood dyscrasias, immunodeficiency, diabetes, among others), who contraindicate the surgical procedure;
* Patients who use medications that interfere with wound healing;
* Pregnant or lactating patients;
* Patients who present opportunistic oral lesions, mainly colonizing the palate region;
* Smoking patients;
* Patients undergoing orthodontic treatment;
* Patients already submitted to periodontal surgery in the area of interest in the present study;
* Patients with a history of allergy to any type of material used in the present study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-21 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Remaining Wound Area (RWA) | baseline, 7, 14, 21, 30, 45 and 90 days after surgery
  For this, standardized photographs will be taken. As a reference, a scale will be used to measure this area. These photographs will be exported to image software (Image J - National Institute of Health -NIH, Bethesda, USA), the area of the wound will be measured in square millimeters (Dias et al. 2015)

SECONDARY OUTCOMES:
Tissue Thickness | baseline, 45 and 90 days after the procedure
  An endodontic spacer (Dentsply-Maillefer Instruments S.A. - Switzerland) with a rubber cursor will be placed in contact with the area until the palatal bone is reached, without pressing the tissue. The distance between the tip of the spacer and the cursor will be measured using a digital caliper (Dias et al., 2015).
Scar and Tissue Colorimetry | 7, 14, 21, 30, 45 and 90 postoperative days
  The presence or absence of scar or keloid in the operated area will be analyzed. In addition, the tissue color similarity of regions adjacent to the operated area and postoperative images will be analyzed through photographs. The photographs will be exported to image software (Adobe Photoshop, München, Germany), using two areas, the wound and one adjacent. The comparison (ΔE) of the areas will be made using brightness parameters (L), red-green chroma scale and blue-yellow chroma scale (b) according to the following equation (Knösel et al., 2009): ΔE =[(L.wound - L.adjacent)2 + (a.wound - a.adjacent)2 + (b.wound - b.adjacent)2] 1/ 2
Epithelialization | baseline, 3, 7, 14 and 30 days after the procedure
  The wound will be colored with Shirley's solution and the epithelialized area will be quantified in the Image J. program. Then, with the total wound area, the % epithelialization will be calculated (Ozcelik et al., 2008).
Early wound healing index | 7 and 14 days after surgery
  Any changes in wound healing will be evaluated, with five different degrees:
  * Complete wound closure with absence of fibrin on the palate;
  * Complete wound closure with the presence of a fibrin line on the palate;
  * Complete wound closure with the presence of a fibrin clot on the palate;
  * Incomplete wound closure with partial tissue necrosis on the palate;
  * Incomplete wound closure with total tissue necrosis on the palate.
Tissue edema | 7 days after the surgical procedure
  It will be evaluated with the score: 1 = absent; 2 = slight; 3 = moderate; or 4 = severe (Sanz-Moliner et al. 2013).
Postoperative discomfort | 7, 14, 21, 30, 45 and 90 days after the surgical procedure
  Sensitivity will be measured by air spray for 5 s over the palatal region. After the air spray, patients will be required to use a 100 mm visual analog scale (VAS) to assess discomfort, where the extremes of the scale will be "none" and "extreme" to report the discomfort of this measure (Dias et al. 2015)
Number of analgesics | until 14 days after surgery
  Patients will be given a postoperative diary in which they will note their pain intensity on a visual analog scale (VAS) 100 mm and the number of painkillers used (Tonetti et. al 2017).
Immunologic Analysis - cytokines | 3 and 7 days after surgery
  The inflammatory exudate present in the palate open wound region will be collected. Samples will be obtained by placing strips of filter paper for 40 s (PerioPaper, Oraflow, New York, USA) in contact with the open wound. After the volume measurements (Periotron 8000, Oraflow, New York, USA), the strips will be placed in sterile tubes containing 300 ml of phosphate buffered saline (PBS) with 0.05% Tween-2 and stored immediately at -80 ° C. Strips contaminated with visible blood will be discarded. The following cytokines will be evaluated: Interleukin-1β (IL1β), Interleukin-4 (IL4), Interleukin-5 (IL5), Interleukin-6 (IL6), Interleukin-9 (IL9), Interleukin-10 (IL10), Interleukin-17A (IL17A), and tumor necrosis factor alpha (TNFα).
Immunologic Analysis - growth factors | 3 and 7 days after surgery
  The inflammatory exudate present in the palate open wound region will be collected. Samples will be obtained by placing strips of filter paper for 40 s (PerioPaper, Oraflow, New York, USA) in contact with the open wound. After the volume measurements (Periotron 8000, Oraflow, New York, USA), the strips will be placed in sterile tubes containing 300 ml of phosphate buffered saline (PBS) with 0.05% Tween-2 and stored immediately at -80 ° C. Strips contaminated with visible blood will be discarded. The following growth factors will be evaluated: Epidermal growth factor (EGF), Transforming growth factor beta (TGF-β), Platelet-derived growth factor (PDGF), Fibroblast growth factors (FGF), and Vascular endothelial growth factor (VEGF).
Immunologic Analysis - matrix metalloproteinases | 3 and 7 days after surgery
  The inflammatory exudate present in the palate open wound region will be collected. Samples will be obtained by placing strips of filter paper for 40 s (PerioPaper, Oraflow, New York, USA) in contact with the open wound. After the volume measurements (Periotron 8000, Oraflow, New York, USA), the strips will be placed in sterile tubes containing 300 ml of phosphate buffered saline (PBS) with 0.05% Tween-2 and stored immediately at -80 ° C. Strips contaminated with visible blood will be discarded. The following Matrix metalloproteinases will be evaluated: matrix metalloproteinase 9 (MMP-9), matrix metalloproteinase 2 (MMP-2), and Tissue inhibitors of metalloproteinases 1 and 2 (TIMP-1/TIMP-2).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, Study Director — Sao Paulo States University - Brazil; Ana Carolina F Bonafe, Principal Investigator — Sao Paulo States University - Brazil
Locations (1):
- Mauro Pedrine Santamaria and Ana Carolina Ferreira Bonafe, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kamalathevan P, Ooi PS, Loo YL. Silk-Based Biomaterials in Cutaneous Wound Healing: A Systematic Review. Adv Skin Wound Care. 2018 Dec;31(12):565-573. doi: 10.1097/01.ASW.0000546233.35130.a9. PMID 30475285
- [Background] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688
- [Background] Zheng Z, Liu Y, Huang W, Mo Y, Lan Y, Guo R, Cheng B. Neurotensin-loaded PLGA/CNC composite nanofiber membranes accelerate diabetic wound healing. Artif Cells Nanomed Biotechnol. 2018;46(sup2):493-501. doi: 10.1080/21691401.2018.1460372. Epub 2018 Apr 13. PMID 29653498
- [Background] Pereira da Silva L, Miguel Neves B, Moura L, Cruz MT, Carvalho E. Neurotensin decreases the proinflammatory status of human skin fibroblasts and increases epidermal growth factor expression. Int J Inflam. 2014;2014:248240. doi: 10.1155/2014/248240. Epub 2014 Aug 11. PMID 25180119